CLINICAL TRIAL: NCT06950580
Title: Investigation of the Effect of Abdominal Massage on Patients in Intensive Care Unit: Randomised Controlled Trial
Brief Title: Effect of Abdominal Massage on Patients in Intensive Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, A. Oguzhan KUCUK, MD, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/10
Record Dates: First submitted 2025-04-09; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Unit Patients; Physiotherapy and Rehabilitation; Abdominal Massage
Keywords: Intensive care unit patients; Physiotherapy and rehabilitation; Abdominal massage; sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Massage Group (Experimental): In addition to routine physiotherapy, patients will receive abdominal massage daily for 5 days.
  Interventions: Other: abdominal massage
- Control Group (No Intervention): Routine physiotherapy will be continued for patients in this group.

INTERVENTIONS:
Other: abdominal massage — In addition to routine physiotherapy, abdominal massage will be applied by the physiotherapist. The patient is positioned supine. The abdominal muscles are stroked three times, followed by colon stroking performed three times, and colon kneading performed three times. The massage is concluded by repeating the colon and abdominal stroking techniques in the same manner. Patients hospitalized in the intensive care unit will routinely receive abdominal massage twice daily by the physiotherapist
  Arms: Abdominal Massage Group

SUMMARY:
Bowel motility can be affected by many factors such as immobilization, lack of fiber in the nutritional formula, inadequate fluid intake, and lack of privacy for toileting in patients hospitalized in the intensive care unit. Abdominal massage, which is one of the effective methods to increase intestinal motility, is accepted as an intervention that can be safely applied in patients.

The aim of our study was to investigate the effect of abdominal massage applied to patients hospitalized in the intensive care unit on sepsis, survival, discharge time from intensive care unit, amount and duration of antibiotic use.

Hypotheses H0: Abdominal massage application has no effect on sepsis, survival, discharge time from intensive care unit, amount and duration of antibiotic use in patients hospitalized in intensive care unit.

H1: Abdominal massage application has an effect on sepsis, survival, discharge time from intensive care unit, amount and duration of antibiotic use in patients hospitalized in intensive care unit.

In this randomized controlled study, the data of patients who received abdominal massage for 5 days during routine physiotherapy applications and those who did not will be recorded. Randomization will be performed in a 1:1 ratio using a computer generated randomization schedule. The effect of abdominal massage on sepsis, survival, discharge time from intensive care, amount and duration of antibiotic use will be examined by using the data of 2 groups with and without abdominal massage in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 80 years
* Patients hospitalized in the intensive care unit for more than 3 days
* Body Mass Index less than 30 kg/m²
* Patients who are not mobilized out of bed
* Patients without any intervention contraindicating abdominal massage

Exclusion Criteria:

* History of abdominal surgery
* Active gastrointestinal bleeding
* Patients discharged from ICU within less than 5 days after enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Sepsis During Follow-Up | From ICU admission through Day 5 of follow-up
  Sepsis will be assessed and recorded according to the Sepsis-3 definition, which requires the presence of suspected or confirmed infection and an acute increase in SOFA (Sequential Organ Failure Assessment) score of ≥2 points from baseline.
  Data for sepsis diagnosis will be collected from daily clinical evaluations, vital signs, laboratory parameters (white blood cell count, procalcitonin, CRP, blood cultures), and organ function assessments. All assessments will be performed by ICU physicians and verified using electronic medical records.
Survival Rate During Follow-Up | From ICU admission through Day 5 of follow-up
  Survival will be assessed by recording the number of patients who remain alive from ICU admission until the end of the 5-day follow-up period.
Length of ICU Stay | From ICU admission through Day 5 of follow-up
  Length of stay in the intensive care unit will be measured in days, calculated as the number of days between the date of ICU admission and the date of ICU discharge. Information will be extracted from patient medical records.
Duration of Antibiotic Use | From ICU admission through Day 5 of follow-up, recorde in days
  The total number of days each patient receives antibiotic treatment will be recorded during the 5-day follow-up period in the ICU. Data will be collected from medication administration records in the patient's medical file.
Amount of Antibiotic Consumption | From ICU admission through Day 5 of follow-up, recorded in milligrams (mg)
  The cumulative amount of antibiotics administered to each patient during the 5-day follow-up period will be recorded in milligrams (mg). Data will be obtained from electronic medication administration records in the ICU.